CLINICAL TRIAL: NCT06277219
Title: A Phase 1/2, Dose-Escalation and Cohort-Expansion Study to Evaluate the Safety, Tolerability, Immunogenicity, Pharmacokinetics, and Efficacy of LAT010 in Patients With Advanced Solid Tumors (LIGHTSPEED-1)
Brief Title: A First-in-Human, Phase 1/2 Study of LAT010 in Patients With Advanced Solid Tumors (LIGHTSPEED-1)
Acronym: LIGHTSPEED-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Latticon Antibody Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LAT010-01
Record Dates: First submitted 2024-02-03; First posted 2024-02-26 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 LAT010 Dose Escalation (Experimental): LAT010 monotherapy with ascending doses in patients with locally advanced or metastatic solid tumors. LAT010 will be administered in planned 7 dose cohorts to determine safety and RP2D. PD profile of LAT010 will also be characterized.
  Interventions: Drug: LAT010
- Phase 2 LAT010 Dose Expansion (Experimental): LAT010 monotherapy at the RP2D and in combination with a PD-1 inhibitor in patients with selected tumor types. LAT010 will be administered at multiple dose levels based on the results of Phase 1. Antitumor activity and safety will be further evaluated.
  Interventions: Drug: LAT010; Drug: LAT010 + ICI

INTERVENTIONS:
Drug: LAT010 — LAT010 monotherapy
Drug: LAT010 + ICI — LAT010 combination with PD-1 inhibitor
  Arms: Phase 2 LAT010 Dose Expansion

SUMMARY:
This is an open-label, multicenter, Phase 1/2, first-in-human (FIH), dose-escalation and cohort-expansion study of LAT010 to evaluate the safety, tolerability, immunogenicity, PK, PD, and antitumor activity in patients with advanced solid tumors. The study consists of 2 parts: Phase 1 dose-escalation and Phase 2 cohort expansion.

DETAILED DESCRIPTION:
Interleukin-2 (IL-2) agonists have shown significant antitumor activities but are associated with severe toxic side effects, due to prioritized activation of high-affinity IL-2 receptor (i.e., IL2Rαβγ). LAT010 is a human IL-2 based immunocytokine designed to exclusively interact with intermediate-affinity IL-2 receptor (i.e., IL2Rβγ) but not the high-affinity IL2Rαβγ receptor. Its exceptional selectivity in activating CD8+ T cells and NK cells may confer the clinical benefits of IL-2 in promoting antitumor immunity without the associated safety concerns.

Phase 1 of the study will examine LAT010 in an accelerated and standard "3+3" dose-escalation design. It consists of 7 planned cohorts. Approximately 20 to 50 patients with locally advanced or metastatic solid tumors will be enrolled in the cohorts. Each treatment cycle consists of 4 weeks, during which patients will receive an IV injection of LAT010 at the assigned dose once weekly. The DLT observation period is the first treatment cycle (28 days).

Phase 2 will be initiated after the MTD or a RP2D has been determined in Phase 1. Approximately up to 30 patients per cohort by tumor type will be enrolled to further evaluate the safety and efficacy of LAT010 in the treatment of selected tumor types at multiple dose levels based on the results of Phase 1. The primary objective of Phase 2 study is to define the preliminary efficacy in the setting of advanced cancers with high unmet medical needs.

ELIGIBILITY:
Inclusion Criteria:

For Phase 1 and Phase 2:

1. Patients have voluntarily signed the informed consent.
2. Patients are willing and able to comply with the protocol-related procedures (including screening evaluations), such as visits, treatment plans, laboratory assessments, and other requirements of the study.
3. Male or female aged ≥18 years old.
4. Patients meet the following diagnoses:

   * Patients have histologically or cytologically documented diagnosis of locally advanced or metastatic solid tumors with evidence of progressive disease according to RECIST 1.1, and
   * Patients are intolerant to or have progressed on all established standard therapies associated with clinical benefit or patients consent that they may be delaying or forgoing treatments known to confer a clinical benefit for their disease, or
   * No additional established line of standard therapy is available, or
   * There is a contraindication for the indicated standard therapies in the opinion of the Investigator.

   (Note: Tumor types of primary interest in Phase 1 include but are not limited to malignant melanoma, renal cell carcinoma, non-small cell lung cancer, gastric carcinoma, hepatocellular carcinoma, pancreatic adenocarcinoma, breast carcinoma, ovarian carcinoma, and colorectal carcinoma.)
5. Patients have at least one measurable tumor lesion, defined as a lesion with the longest measurable diameter of non-lymph node lesions by imaging (CT/MRI) of ≥10 mm or the short diameter of a single pathological lymph node lesion of ≥15 mm.
6. Expected life expectancy of >12 weeks per the Investigator.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 for Phase 1. ECOG score of 0 to 2 for Phase 2.
8. If a patient has had prior major surgery, at least 4 weeks must have elapsed at the time of screening.
9. Patients have adequate pulmonary, cardiovascular, hematological, liver, and renal function, per Investigator assessment.
10. Patients have not received any IL-2 therapy within 12 months before the first dose of LAT010.
11. Laboratory values at screening are as follows:

    a. Hematology: i. Absolute neutrophil count (ANC) ≥1,500 cells/mm3 ii. Platelet count ≥75,000 cells/mm3 (no blood components or cell growth factors are used as supportive care within 7 days before the first dose of LAT010) iii. Hemoglobin ≥9.0 g/dL, transfusion of red blood cells allowed to reach threshold target if >7 days b. Renal: i. Creatinine clearance >30 mL/min as derived from the Cockcroft-Gault glomerular filtration rate estimation c. Coagulation: i. International Normalized Ratio (INR) ≤1.5× the upper limit of normal (ULN) ii. Prothrombin time (PT) or activated partial thromboplastin time (APTT) ≤1.5×ULN unless undergoing anticoagulation therapy d. Liver: i. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3.0×ULN without liver metastasis or ≤5×ULN with liver metastasis ii. Bilirubin <1.5×ULN (unless Gilbert syndrome is confirmed)
12. Any toxicity of previous treatment has recovered to Grade ≤1, unless the toxicity is judged by the Investigator to pose no safety risk, such as alopecia (any grade) or fatigue (up to Grade 2 allowed).
13. Female patients of childbearing potential and sexually active male patients with female partners of childbearing potential must agree to use effective contraceptive measures (including concomitant use of a spermicide with barrier method, intrauterine device, or hormonal contraceptives) from signing the informed consent form to at least 90 days after the last dose of LAT010. Female patients of childbearing age and women <12 months after menopause must have a negative pregnancy test result within 7 days before the first dose of LAT010.
14. Male patients must not donate sperm starting at screening and throughout the study period and for at least 90 days after the final study drug administration.

    For Phase 2 only:
15. Patients must meet the following criteria:

    1. Patients are willing and able to undergo baseline and on-treatment biopsies of the tumor. If a patient has residual tumor masses that can only be accessed with significant risk, available archived biopsies (frozen or formalin-fixed) may serve as baseline specimens with the Sponsor's approval.
    2. Patients have been diagnosed and histologically confirmed with a tumor type being selected for the Phase 2 trial.
    3. Patients have received the established standard therapies for the selected tumor type prior to enrolling to this study and patients consent that they may be delaying or forgoing specific treatments known to confer a clinical benefit for their disease.
    4. Must have received no more than 1 prior line of anti-angiogenic therapy, e.g., anti-vascular endothelial growth factor (anti-VEGF) therapy

Exclusion Criteria:

1. Cardiovascular exclusions:

   1. Patient has a medical history of an arterial thrombotic event, stroke, or transient ischemia attack within the past 6 months.
   2. Patient has a medical history of symptomatic congestive heart failure (New York Heart Association classes III or IV) or an uncontrolled clinically significant cardiac arrhythmia that requires treatment.
   3. Patient has a medical history of myocardial infarction or unstable angina within 6 months before the first dose of LAT010.
   4. Patient has a QTc prolongation to >480 milliseconds (ms) based on a 12-lead ECGs in triplicate.
2. Other exclusions:

   1. Patient is actively enrolled in another clinical study, unless it is an observational (noninterventional) clinical study or the follow-up component of an interventional study.
   2. Use of another systemic anti-cancer therapy within 3 weeks or 5 half- lives after the first dose of LAT010, whichever is shorter.
   3. Patient has active central nervous system (CNS) metastases. However, definitely treated CNS metastases (such as surgery, radiotherapy) that are stable for at least 2 weeks prior to the first dose of LAT010 are acceptable.
   4. Patient has another active primary malignancy that has not been treated with curative intent. Exceptions could be made upon discussion with the Medical Monitor. However, non-metastatic cutaneous basal cell or squamous cell carcinoma, or non-muscle invasive bladder cancer are acceptable.
   5. Patient has history of severe irAEs from a previous treatment, which are defined as a Grade 4 event requiring corticosteroid treatment or a Grade 3 event requiring corticosteroid treatment of >10 mg/day prednisone or equivalent dose for >12 weeks.
3. Recent medical concerns exclusions:

   1. Patient has evidence of active infection requiring IV antibiotics within 7 days prior to the first dose of LAT010.
   2. Patient has active uncontrolled bleeding within 7 days prior to the first dose of LAT010.
   3. Patient has serious or non-healing wound, fistula, skin ulcer, or non-healing bone fracture within 7 days prior to the first dose of LAT010.
   4. Patient has had a live virus vaccine within 30 days prior to the first dose of LAT010 (Note: Inactivated seasonal flu vaccine is acceptable. COVID-19 vaccination is also allowed.)
4. Patient has known replicating human immunodeficiency virus infection, active hepatitis B infection, or hepatitis C infection. However, hepatitis B virus (HBV) carriers without active disease (HBV DNA titer < 1000 cps/mL or 200 IU/mL) or patients with cured hepatitis C (negative HCV RNA test) may be enrolled. Patients with treated non-replicative disease are acceptable.
5. Patient is taking corticosteroids >10 mg/day of prednisone or equivalent.
6. Patient has had an organ transplantation or is on systemic immunosuppressive therapy.
7. Patient has a positive test result for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) viral RNA test, either asymptomatic or present with symptoms of Coronavirus disease 2019 (COVID-19) on Day -2 or Day -1.
8. Patient has a serious illness considered by the Investigator to be unsuitable for participating in this study.
9. Any condition that, in the opinion of the Investigator, may interfere with the evaluation of the study drug or interpretation of the patient's safety or study results.
10. Patient has a history of sensitivity to LAT010, or components thereof, or a history of drug or other allergy that in the opinion of the Investigator or Medical Monitor (if appropriate), contraindicates their participation.
11. Patient has any illness, medical condition, organ system dysfunction, or social situation, including mental illness or substance abuse, that is deemed by the Investigator to be likely to interfere with a patient's ability to sign the informed consent form (ICF), adversely affect the patient's ability to cooperate and participate in the study, or compromise the interpretation of study results.
12. Patient is breastfeeding or pregnant as confirmed by pregnancy tests performed within 7 days before the first dose of LAT010.
13. Patient is unwilling or unable to follow protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) (Phase 1) | Up to 18 months
  TEAEs
Incidence of changes in clinical laboratory values (Phase 1) | Up to 15 months
  Clinical Lab Values
Incidence of dose-limiting toxicities (DLTs) (Phase 1) | The first treatment cycle (28 days) from Cycle 1 Day 1
  DLT
Objective response rate (ORR) per RECIST 1.1 (Phase 2) | Up to 24 months
  ORR

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of LAT010 | Through treatment cycles, up to approximately 1 year
  Cmax
Area under the plasma concentration-time curve (AUC) of LAT010 | Through treatment cycles, up to approximately 1 year
  AUC
Terminal phase half-life (t1/2) of LAT010 | Through treatment cycles, up to approximately 1 year
  t½
Time to maximum concentration of LAT010 | Through treatment cycles, up to approximately 1 year
  Tmax
Trough concentration of LAT010 | Through treatment cycles, up to approximately 1 year
  Ctrough
Volume of distribution of LAT010 | Through treatment cycles, up to approximately 1 year
  Vd
Clearance of LAT010 | Through treatment cycles, up to approximately 1 year
  CL
ADA occurrence and titer in serum | Through safety follow-up period, up to approximately 15 months
  ADA
Objective response rate (ORR) per RECIST 1.1 (Phase 1 ) | Up to 24 months
  ORR
Duration of response (DOR) | Up to 24 months
  DOR
Disease control rate (DCR) | Up to 24 months
  DCR
Progression-free survival (PFS) | Up to 24 months
  PFS
Overall survival (OS) | Up to 24 months
  OS
Incidence of AEs and SAEs | From informed consent signed through safety follow-up period, up to approximately 15 months
  AEs/SAEs

OTHER OUTCOMES:
Epigenetic assessment of the proliferation and activation of CD4+ Treg cells, CD8+ T cells, and natural killer (NK) cells. | Through the end of Cycle 1 (each cycle is 28 days) in Phase 1
  PD
Optional flow cytometry assessment of the proliferation and activation of CD4+ Treg cells, CD8+ T cells, and NK cells. | Through treatment cycles in Phase 2, up to approximately 1 year
  PD

CONTACTS AND LOCATIONS:
Overall Officials: John Li, PhD, Study Chair — Latticon Antibody Therapeutics, Inc
Locations (4):
- United States (2):
  - D&H Cancer Research Center, Margate, Florida
  - Huntsman Cancer Institute, Salt Lake City, Utah
- China (2):
  - Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No